CLINICAL TRIAL: NCT00005303
Title: Effectiveness of AIDS Antibody Screening
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 3004
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: Acquired Immunodeficiency Syndrome; Blood Transfusion; HIV Infections
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections

STUDY DESIGN:
Observational Model: Natural History

SUMMARY:
To determine the effectiveness of efforts to eliminate the human immunodeficiency virus (HIV) from whole blood and blood components in the blood supply.

DETAILED DESCRIPTION:
BACKGROUND:

In 1986, despite programs to have persons with known risk factors for exposure to the AIDS virus exclude themselves from the blood donating population and the universal testing of all donated whole blood and blood components for the antibody to HIV, the public was fearful of acquiring AIDS via transfusion and media stories increased that fear. A major concern among members of the blood banking community was the extent to which donors infected with HIV were not identified by enzyme-linked immunoassay (EIA) systems. Most experts believed that self-deferral and the assays for the HIV antibody were eliminating the vast majority of positive units of donated blood and blood components. If all units containing HIV were being eliminated by the combined effects of self-deferral and antibody screening (and treatment of factor VIII concentrates), no recipients of only screened whole blood or blood components or factor VIII would become HIV virus and antibody positive as the result of transfusion. Alternately, if some HIV positive units of whole blood or blood components or factor VIII concentrates were not being eliminated by self-deferral and antibody screening (and treatment of factor VIII concentrates), and these units were transfused, then some transfusion recipients would become HIV antibody positive and viremic.

The initiative was part of a special Fiscal Year 1986 National Heart, Lung, and Blood Institute AIDS Plan. The concept was reviewed and approved by the National Heart, Lung, and Blood Advisory Council in February 1986. The Request for Proposals was released in May 1986. Two contracts were awarded in September 1986.

DESIGN NARRATIVE:

University of California at San Francisco: A risk assessment was made of HIV infection through prospective testing for seroconversion in women recipients of anti-HIV negative blood transfusions at the University of California San Francisco hospitals. Blood specimens were collected from each of the recipients pre-transfusion, and at two, four, and six months post-transfusion. Patients were selected based on female sex and exclusion of high risk behavior or blood transfusion during the preceding six months.

Johns Hopkins University: The rate of seroconversion was determined in a cohort of cardiac surgery patients receiving multiple transfusions of blood products screened for HIV antibody. The study was conducted at the Johns Hopkins Hospital, the Texas Heart Institute, and the Methodist Hospital in Houston. A serum sample for each patient was collected before surgery and a second sample was collected at least six months after surgery.

ELIGIBILITY:
No eligibility criteria

Min Age: 0 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1986-09; Study Completion 1995-09

CONTACTS AND LOCATIONS:
Overall Officials: Girish Vyas

REFERENCES:
- [Background] Ulrich PP, Busch MP, el-Beik T, Shiota J, Vennari J, Shriver K, Vyas GN. Assessment of human immunodeficiency virus expression in cocultures of peripheral blood mononuclear cells from healthy seropositive subjects. J Med Virol. 1988 May;25(1):1-10. doi: 10.1002/jmv.1890250102. PMID 3411308
- [Background] Hwang LY, Beasley RP, Busch MP, Lane PK, Vyas GN. Human immunodeficiency virus seroprevalence among blood product recipients in San Francisco before transfusion. Transfusion. 1989 Feb;29(2):113-8. doi: 10.1046/j.1537-2995.1989.29289146827.x. PMID 2919421
- [Background] Scillian JJ, McHugh TM, Busch MP, Tam M, Fulwyler MJ, Chien DY, Vyas GN. Early detection of antibodies against rDNA-produced HIV proteins with a flow cytometric assay. Blood. 1989 May 15;73(7):2041-8. PMID 2540862
- [Background] Roy S, Morrow WJ, Christian C, Khayam-Bashi H, Busch MP, McCarthy R, Rodgers RP, Vyas GN. Persistent immune complexes and abnormal CD4/CD8 ratios in HIV infection. J Acquir Immune Defic Syndr (1988). 1990;3(2):134-8. PMID 1967308
- [Background] Cohen ND, Munoz A, Reitz BA, Ness PK, Frazier OH, Yawn DH, Lee H, Blattner W, Donahue JG, Nelson KE, et al. Transmission of retroviruses by transfusion of screened blood in patients undergoing cardiac surgery. N Engl J Med. 1989 May 4;320(18):1172-6. doi: 10.1056/NEJM198905043201803. PMID 2710190
- [Background] Yang G, Olson JC, Pu R, Vyas GN. Flow cytometric detection of human immunodeficiency virus type 1 proviral DNA by the polymerase chain reaction incorporating digoxigenin- or fluorescein-labeled dUTP. Cytometry. 1995 Oct 1;21(2):197-202. doi: 10.1002/cyto.990210212. PMID 8582240
- [Background] Yang G, Garhwal S, Olson JC, Vyas GN. Flow cytometric immunodetection of human immunodeficiency virus type 1 proviral DNA by heminested PCR and digoxigenin-labeled probes. Clin Diagn Lab Immunol. 1994 Jan;1(1):26-31. doi: 10.1128/cdli.1.1.26-31.1994. PMID 7496917
- [Background] Babu PG, Rawal BD, Khayam-Bashi H, Vyas GN. Detection of exceedingly low levels of HIV proviral DNA in multimillion peripheral blood mononuclear cells by PCR. PCR Methods Appl. 1993 Aug;3(1):63-4. doi: 10.1101/gr.3.1.63. No abstract available. PMID 8220187
- [Background] Yang G, Ulrich PP, Aiyer RA, Rawal BD, Vyas GN. Detection of hepatitis B virus in plasma using flow cytometric analyses of polymerase chain reaction-amplified DNA incorporating digoxigenin-11-dUTP. Blood. 1993 Feb 15;81(4):1083-8. PMID 8427989
- [Background] Busch MP, Eble BE, Khayam-Bashi H, Heilbron D, Murphy EL, Kwok S, Sninsky J, Perkins HA, Vyas GN. Evaluation of screened blood donations for human immunodeficiency virus type 1 infection by culture and DNA amplification of pooled cells. N Engl J Med. 1991 Jul 4;325(1):1-5. doi: 10.1056/NEJM199107043250101. PMID 2046708
- [Background] Donahue JG, Munoz A, Ness PM, Brown DE Jr, Yawn DH, McAllister HA Jr, Reitz BA, Nelson KE. The declining risk of post-transfusion hepatitis C virus infection. N Engl J Med. 1992 Aug 6;327(6):369-73. doi: 10.1056/NEJM199208063270601. PMID 1320736
- [Background] Nelson KE, Donahue JG, Munoz A, Cohen ND, Ness PM, Teague A, Stambolis VA, Yawn DH, Callicott B, McAllister H, et al. Transmission of retroviruses from seronegative donors by transfusion during cardiac surgery. A multicenter study of HIV-1 and HTLV-I/II infections. Ann Intern Med. 1992 Oct 1;117(7):554-9. doi: 10.7326/0003-4819-117-7-554. PMID 1524329
- [Background] Donahue JG, Nelson KE, Munoz A, Vlahov D, Rennie LL, Taylor EL, Saah AJ, Cohn S, Odaka NJ, Farzadegan H. Antibody to hepatitis C virus among cardiac surgery patients, homosexual men, and intravenous drug users in Baltimore, Maryland. Am J Epidemiol. 1991 Nov 15;134(10):1206-11. doi: 10.1093/oxfordjournals.aje.a116023. PMID 1720924